CLINICAL TRIAL: NCT02675114
Title: A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients Who Have Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: PARTNER 3 Trial: Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients With Aortic Stenosis
Acronym: P3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-08
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Aortic Stenosis
Keywords: SAPIEN 3; cardiovascular disease; heart disease; aortic stenosis; Surgical aortic valve replacement (SAVR); Transcatheter aortic valve replacement (TAVR)
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Surgical aortic valve replacement (SAVR) (Active Comparator)
  Interventions: Procedure: SAVR
- Transcatheter aortic valve replacement (TAVR) (Experimental)
  Interventions: Device: SAPIEN 3 THV

INTERVENTIONS:
Procedure: SAVR — SAVR with a commercially available bioprosthetic valve.
  Arms: Surgical aortic valve replacement (SAVR)
Device: SAPIEN 3 THV — TAVR with the Edwards SAPIEN 3 Transcatheter Heart Valve and Edwards Commander Delivery System
  Arms: Transcatheter aortic valve replacement (TAVR)

SUMMARY:
To establish the safety and effectiveness of the Edwards SAPIEN 3 Transcatheter Heart Valve (THV) in patients with severe, calcific aortic stenosis who are at low operative risk for standard aortic valve replacement.

DETAILED DESCRIPTION:
Prospective, randomized, controlled, multi-center trial. Patients having an operative mortality < 4% (low operative risk) for surgical aortic valve replacement will be randomized 1:1 to receive either transcatheter heart valve replacement (TAVR) with the Edwards SAPIEN 3 or aortic valve replacement with a commercially available surgical bioprosthetic valve. Patients will be seen for follow-up visits at discharge, 30 days, 6 months, and annually through 10 years.

A subset of PARTNER 3 randomized patients will be enrolled in the Actigraphy/Quality of Life. Additional patients will be enrolled in either the Bicuspid Registry, Underrepresented Populations Registry (UPR) or the Alternative Access Registry.

ELIGIBILITY:
Inclusion Criteria:

1. Severe, calcific aortic stenosis
2. New York Heart Association Functional Class ≥ 2 OR exercise tolerance test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR asymptomatic with Left Ventricular Ejection Fraction (LVEF) <50%
3. Heart team agrees the patient has a risk of operative mortality and has an Society of Thoracic Surgeons (STS) score < 4
4. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Native aortic annulus size unsuitable for sizes 20, 23, 26, or 29 mm transcatheter heart valve
2. Iliofemoral vessel characteristics that would preclude safe passage of the introducer sheath
3. Evidence of an acute myocardial infarction ≤ 30 days before randomization
4. Aortic valve is unicuspid, bicuspid, or non-calcified
5. Severe aortic regurgitation (>3+)
6. Severe mitral regurgitation (>3+) ≥ moderate stenosis
7. Pre-existing mechanical or bioprosthetic valve in any position
8. Complex coronary artery disease:

   1. Unprotected left main coronary artery
   2. Syntax score > 32
   3. Heart Team assessment that optimal revascularization cannot be performed
9. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of randomization
10. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy, or hypercoagulable states
11. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of randomization
12. Hypertrophic cardiomyopathy with obstruction
13. Ventricular dysfunction with LVEF < 30%
14. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
15. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure
16. Stroke or transient ischemic attack within 90 days of randomization
17. Renal insufficiency and/or renal replacement therapy at the time of screening.
18. Active bacterial endocarditis within 180 days of randomization
19. Severe lung disease or currently on home oxygen
20. Severe pulmonary hypertension
21. History of cirrhosis or any active liver disease
22. Significant frailty as determined by the Heart Team
23. Significant abdominal or thoracic aortic disease that would preclude safe passage of the delivery system or cannulation and aortotomy for surgical aortic valve replacement
24. Hostile chest or conditions or complications from prior surgery that would preclude safe reoperation
25. Patient refuses blood products
26. Body mass index > 50 kg/m2
27. Estimated life expectancy < 24 months
28. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
29. Immobility that would prevent completion of study procedures
30. Patient is not a candidate for both arms of the study
31. Currently participating in an investigational drug or another device study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, FACC, Principal Investigator — Columbia University Medical Center/ New York Presbyterian Hospital, NY; Michael J Mack, MD, FACC, Principal Investigator — The Heart Hospital Baylor Plano, TX
Locations (77):
- United States (68):
  - University of Alabama, Birmingham, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - Mills/Peninsula Health Services, Burlingame, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles/Ronald Reagan Medical Center, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Sutter Health Sacramento, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - UC Health Northern Colorado/Medical Center of the Rockies, Loveland, Colorado
  - Hartford, Hartford, Connecticut
  - JFK Medical Center / Atlantic Clinical Research Collaborative, Atlantis, Florida
  - University of Florida, Gainesville, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem Research Institute, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - UPR - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Central Maine Medical Center, Auburn, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - Barnes-Jewish Hospital / Washington University, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Medical Center / Atlantic Health System Hospital, Morristown, New Jersey
  - Newark Beth Israel, Newark, New Jersey
  - Albany, Albany, New York
  - University of Buffalo, Buffalo, New York
  - Winthrop-University Hospital, Mineola, New York
  - NYU Medical Center, New York, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - Carolina's Health System, Charlotte, North Carolina
  - UPR - Novant Health Heart and Vascular Institution, Charlotte, North Carolina
  - Rex Hospital / NC Heart and Vascular Research, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel Health System, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - UPR-Oklahoma Heart Institute, Tulsa, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Saint Thomas Health Services, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hosptial Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Fairfax INOVA, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
- Saint Paul's Hospital, Vancouver, Canada
- Japan (5):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Osaka University, Suita, Osaka
  - Keio University, Shinjuku, Tokyo
  - Teikyo University, tabashi City, Tokyo
- Auckland City Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leon MB, Mack MJ, Pibarot P, Hahn RT, Thourani VH, Kodali SH, Genereux P, Kapadia SR, Cohen DJ, Pocock SJ, Zhang Y, Szerlip M, Ternacle J, Malaisrie SC, Herrmann HC, Szeto WY, Russo MJ, Babaliaros V, Nazif T, Webb JG, Makkar RR; PARTNER 3 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Low-Risk Patients at 7 Years. N Engl J Med. 2025 Oct 27. doi: 10.1056/NEJMoa2509766. Online ahead of print. PMID 41144631
- [Derived] Hahn RT, Ternacle J, Silva I, Giuliani C, Zanuttini A, Theron A, Cristell N, Bernier M, Skaf S, Beaudoin J, Kodali SK, Russo M, Kapadia SR, Malaisrie CS, Cohen DJ, Leipsic J, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Park B, Gunnarsson M, Webb JG, Smith CR, Makkar R, Thourani VH, Mack MJ, Leon MB, Pibarot P; PARTNER 3 Investigators. 5-Year Echocardiographic Results of Transcatheter Versus Surgical Aortic Valve Replacement in Low-Risk Patients. JACC Cardiovasc Imaging. 2025 Jun;18(6):625-640. doi: 10.1016/j.jcmg.2025.01.015. Epub 2025 Apr 16. PMID 40243974
- [Derived] Mack MJ, Leon MB, Thourani VH, Pibarot P, Hahn RT, Genereux P, Kodali SK, Kapadia SR, Cohen DJ, Pocock SJ, Lu M, White R, Szerlip M, Ternacle J, Malaisrie SC, Herrmann HC, Szeto WY, Russo MJ, Babaliaros V, Smith CR, Blanke P, Webb JG, Makkar R; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement in Low-Risk Patients at Five Years. N Engl J Med. 2023 Nov 23;389(21):1949-1960. doi: 10.1056/NEJMoa2307447. Epub 2023 Oct 24. PMID 37874020
- [Derived] Genereux P, Cohen DJ, Pibarot P, Redfors B, Bax JJ, Zhao Y, Prince H, Makkar RR, Kapadia S, Thourani VH, Mack MJ, Nazif TM, Lindman BR, Babaliaros V, Russo M, McCabe JM, Gillam LD, Alu MC, Hahn RT, Webb JG, Leon MB, Arnold SV. Cardiac Damage and Quality of Life After Aortic Valve Replacement in the PARTNER Trials. J Am Coll Cardiol. 2023 Feb 28;81(8):743-752. doi: 10.1016/j.jacc.2022.11.059. PMID 36813373
- [Derived] Kuck KH, Leidl R, Frankenstein L, Wahlers T, Sarmah A, Candolfi P, Shore J, Green M. Cost-Effectiveness of SAPIEN 3 Transcatheter Aortic Valve Implantation Versus Surgical Aortic Valve Replacement in German Severe Aortic Stenosis Patients at Low Surgical Mortality Risk. Adv Ther. 2023 Mar;40(3):1031-1046. doi: 10.1007/s12325-022-02392-y. Epub 2023 Jan 9. PMID 36622552
- [Derived] Genereux P, Pibarot P, Redfors B, Bax JJ, Zhao Y, Makkar RR, Kapadia S, Thourani VH, Mack MJ, Nazif TM, Lindman BR, Babaliaros V, Vincent F, Russo M, McCabe JM, Gillam LD, Alu MC, Hahn RT, Webb JG, Leon MB, Cohen DJ. Evolution and Prognostic Impact of Cardiac Damage After Aortic Valve Replacement. J Am Coll Cardiol. 2022 Aug 23;80(8):783-800. doi: 10.1016/j.jacc.2022.05.006. Epub 2022 May 17. PMID 35595203
- [Derived] Ternacle J, Al-Azizi K, Szerlip M, Potluri S, Hamandi M, Blanke P, Leipsic J, Dahou A, Salaun E, Vincent F, Rogers E, Alu MC, Lu M, Yu X, Thourani VH, Hahn RT, Leon MB, Pibarot P, Mack MJ. Impact of Predilation During Transcatheter Aortic Valve Replacement: Insights From the PARTNER 3 Trial. Circ Cardiovasc Interv. 2021 Jul;14(7):e010336. doi: 10.1161/CIRCINTERVENTIONS.120.010336. Epub 2021 Jun 18. PMID 34139864
- [Derived] Herrmann HC, Cohen DJ, Hahn RT, Babaliaros VC, Yu X, Makkar R, McCabe J, Szerlip M, Kapadia S, Russo M, Malaisrie SC, Webb JG, Szeto WY, Kodali S, Thourani VH, Mack MJ, Leon MB. Utilization, Costs, and Outcomes of Conscious Sedation Versus General Anesthesia for Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2021 Jul;14(7):e010310. doi: 10.1161/CIRCINTERVENTIONS.120.010310. Epub 2021 Jun 16. PMID 34130476
- [Derived] Leon MB, Mack MJ, Hahn RT, Thourani VH, Makkar R, Kodali SK, Alu MC, Madhavan MV, Chau KH, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Blanke P, Leipsic JA, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Herrmann HC, Szeto WY, Genereux P, Pershad A, Lu M, Webb JG, Smith CR, Pibarot P; PARTNER 3 Investigators. Outcomes 2 Years After Transcatheter Aortic Valve Replacement in Patients at Low Surgical Risk. J Am Coll Cardiol. 2021 Mar 9;77(9):1149-1161. doi: 10.1016/j.jacc.2020.12.052. PMID 33663731
- [Derived] Pibarot P, Salaun E, Dahou A, Avenatti E, Guzzetti E, Annabi MS, Toubal O, Bernier M, Beaudoin J, Ong G, Ternacle J, Krapf L, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Leipsic J, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Alu MC, Xu K, Rogers E, Webb JG, Smith CR, Mack MJ, Leon MB, Hahn RT; PARTNER 3 Investigators. Echocardiographic Results of Transcatheter Versus Surgical Aortic Valve Replacement in Low-Risk Patients: The PARTNER 3 Trial. Circulation. 2020 May 12;141(19):1527-1537. doi: 10.1161/CIRCULATIONAHA.119.044574. Epub 2020 Apr 10. PMID 32272848
- [Derived] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Derived] Leipsic J, Bax JJ, Webb JG, Martin R, Blanke P. Trials Testing the Value of Imaging Use in Valve Disease and in Transcatheter Valvular Interventions. JACC Cardiovasc Imaging. 2017 Mar;10(3):286-295. doi: 10.1016/j.jcmg.2016.09.031. PMID 28279376

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Aortic Valve Replacement (SAVR): SAVR with a commercially available bioprosthetic valve.
- Transcatheter Aortic Valve Replacement (TAVR): TAVR with the Edwards SAPIEN 3 Transcatheter Heart Valve and Edwards Commander Delivery System
Period: Overall Study
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Started | 497 | 503
As Treated | 454 | 496
Valve Implant | 453 | 495
Completed | 424 | 490
Not Completed | 73 | 13

BASELINE CHARACTERISTICS:
Population: As Treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR) | Total
Number analyzed (Participants) | 454 | 496 | 950
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.08) | 73.3 (5.83) | 73.4 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 161 | 292
  Male | 323 | 335 | 658
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 8 | 17
  Black or African American | 12 | 15 | 27
  Hispanic or Latino | 9 | 7 | 16
  Native Hawaiian or other Pacific Islander | 4 | 5 | 9
  White | 409 | 458 | 867
  Multiple | 6 | 3 | 9
  Other | 4 | 0 | 4
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality, All Stroke, and Rehospitalization (Valve-related or Procedure-related and Including Heart Failure)
Description: Number of patients that had any of these events
Time Frame: 1 year
Population: As Treated
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 454 | 496
Participants | 68 | 42

2. Secondary Outcome: New Onset Atrial Fibrillation
Description: Number of patients with this event
Time Frame: 30 days
Population: As Treated. Patients who had atrial fibrillation prior to the procedure were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 369 | 417
Participants | 145 | 21

3. Secondary Outcome: Length of Index Hospitalization
Description: Number of days from index procedure to discharge
Time Frame: Discharge (expected average of 7 days)
Population: As Treated
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 454 | 496
Days | 7.4 (3.48) | 2.9 (2.24)

4. Secondary Outcome: Death, Kansas City Cardiomyopathy Questionnaire (KCCQ) Score < 45 or KCCQ Score Decrease ≥ 10 Points
Description: Number of patients that had any of these events
Time Frame: 30 days
Population: As Treated
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 435 | 492
Participants | 133 | 19

5. Secondary Outcome: Death or Stroke
Description: Number of patients that died or had a stroke
Time Frame: 30 days
Population: As Treated
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 454 | 496
Participants | 15 | 5

6. Secondary Outcome: All Stroke
Description: Number of patients that had a stroke
Time Frame: 30 days
Population: As Treated
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
Number analyzed (Participants) | 454 | 496
Participants | 11 | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Surgical Aortic Valve Replacement (SAVR) | Transcatheter Aortic Valve Replacement (TAVR)
All-Cause Mortality (participants affected / at risk) | 11/454 | 5/496
Serious Adverse Events (participants affected / at risk) | 221/454 | 153/496
Other Adverse Events (participants affected / at risk) | 305/454 | 133/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Aortic Valve Replacement (SAVR) (N=454) | Transcatheter Aortic Valve Replacement (TAVR) (N=496)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 9 (9) | 3 (3)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 4 (4) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 4 (4) | 4 (4)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 42 (43) | 11 (12)
Atrial flutter (Cardiac disorders) | 12 (13) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 15 (15) | 22 (23)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 12 (12)
Cardiac arrest (Cardiac disorders) | 5 (6) | 4 (4)
Cardiac failure (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (7) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular enlargement (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Paravalvular aortic regurgitation (Cardiac disorders) | 2 (2) | 4 (4)
Pericardial effusion (Cardiac disorders) | 6 (6) | 2 (2)
Pericardial haemorrhage (Cardiac disorders) | 8 (8) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Systolic anterior motion of mitral valve (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 5 (5) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 10 (11)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oroantral fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Serratia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 13 (14) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Pulmonary arterial pressure increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 7 (7) | 4 (4)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal haematocoele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 2 (2)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericardial excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 2 (2)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Femoral artery dissection (Vascular disorders) | 0 (0) | 3 (3)
Femoral artery perforation (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 3 (3)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 2 (2)
Renovascular hypertension (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Vessel perforation (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Aortic Valve Replacement (SAVR) (N=454) | Transcatheter Aortic Valve Replacement (TAVR) (N=496)
Anaemia (Blood and lymphatic system disorders) | 28 (29) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 59 (60) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (24) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 145 (154) | 36 (38)
Atrioventricular block first degree (Cardiac disorders) | 26 (26) | 26 (26)
Bundle branch block left (Cardiac disorders) | 37 (37) | 92 (93)
Bundle branch block right (Cardiac disorders) | 28 (28) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 88 (89) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 40 (41) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 39 (40) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02675114/Prot_SAP_000.pdf